CLINICAL TRIAL: NCT05985928
Title: Sensory Study: Taste and Tongue Biology
Acronym: SweetTaste
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2587; R21DC018906 (NIH)
Record Dates: First submitted 2023-07-13; First posted 2023-08-14 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2023-05

CONDITIONS: Healthy Adults
Keywords: sweet; genetics; gene expression; dietary intake; psychophysics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — saliva, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Researchers will investigate the correlation between a) self-reported dietary intake of foods and beverages, b) intensity of sucrose stimuli, and c) liking rating of sweet stimuli, with the relative expression of the taste receptor genes from human fungiform papillae (TAS1R2 and TAS1R3).

* This research will provide new information on how sweet taste perception is regulated.

* The hypothesis: Greater dietary consumption of sugar and sweet foods is associated with reduced expression of the sweet taste receptors.
* The results of this study could help to identify pathways to help modify sweet taste perception by uncovering this mechanism.

Participants will sample solutions prepared with sweet ingredients, provide salivary DNA, and collect fungiform papillae. This will allow researchers and investigators to compare the relationship between the sweetness of stimuli, genetic differences in sweet taste receptors, and expression levels of sweet taste receptor genes.

ELIGIBILITY:
Inclusion Criteria:

1. between 18 and 45 years old,
2. have no tongue or cheek piercings,
3. not a user of tobacco products or electronic cigarettes (within the last year),
4. no known defects in taste or smell,
5. not pregnant or breastfeeding,
6. no history of chronic pain in the mouth,
7. not taking any prescription pain medication,
8. not taking any blood thinners,
9. no history of cancer or cancer treatment,
10. not diabetic or restricting intake of sugars for medical reasons, under the direction of a physician or healthcare provider
11. willing to undergo the Fungiform Papillae biopsy procedure
12. willing to provide salivary DNA
13. Not currently experiencing any COVID-19 symptoms
14. Not recently diagnosed (in the last 30 days) with COVID-19
15. No history of high blood pressure

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy adults, over the age of 18, able to provide consent in English, able to complete survey on an electronic device
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Gene expression and sweet taste perception | Day 1 (single time-point)
  The relative level of gene expression of sweet taste receptors (TAS1R2 and TAS1R3) and relationship with sweet taste perception (gLMS ratings of sampled sucrose)
Gene expression and sweet taste liking | Day 1 (single time-point)
  The relative level of gene expression of sweet taste receptors (TAS1R2 and TAS1R3) and relationship with sweet taste perception (hedonic ratings of sampled sucrose)
Gene expression and dietary intake | Day 1 (single time-point)
  The relative gene level expression of sweet taste receptors and relationship with self-reported dietary intake of sweet foods and beverages
Gene expression and sweet liker status | Day 1 (single time-point)
  The relative gene level expression of sweet taste receptors and relationship with the self-reported liking of a variety of sweet foods and beverages

SECONDARY OUTCOMES:
Genetics and sweet taste perception | Day 1 (single time-point)
  Genetic variability in sweet taste receptor genes and the relationship with perception of sweet stimuli (gLMS intensity ratings)
Genetics and sweet taste liking | Day 1 (single time-point)
  Genetic variability in sweet taste receptor genes and the relationship with hedonic ratings of sweet stimuli (hedonic ratings)
Genetics and sweet liker status | Day 1 (single time-point)
  Genetic variability in sweet taste receptor genes and the relationship with the self-reported liking of sweet-tasting foods and beverages

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared at the request, after signing release form. No PHI will be included. All data will be de-identified. Data and meta-data will be shared, along with code books.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available following publication of results.
Access Criteria: Individuals can access the following signing form from IRB.